CLINICAL TRIAL: NCT03450850
Title: Phase II, Single Arm Study Of NOVOTTF-200A In Bevacizumab-Naive Subjects With Recurrent WHO Grade III Malignant Astrocytoma
Brief Title: Study Of NOVOTTF-200A In Bevacizumab-Naive Subjects With Recurrent Grade III Malignant Astrocytoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela A. Bota (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Daniela A. Bota, Associate Professor, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20174031; UCI 16-56 (Other: UCI CFCCC)
Record Dates: First submitted 2018-01-23; First posted 2018-03-01 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Astrocytoma, Grade III
MeSH Terms: conditions — Astrocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NOVOTTF-200A (Other): NOVOTTF-200A treatment in Bevacizumab-Naïve Subjects with Recurrent WHO Grade III Malignant Astrocytoma
  Interventions: Device: NOVOTTF-200A

INTERVENTIONS:
Device: NOVOTTF-200A — NOVOTTF-200A will be administered under appropriate guidelines. Monthly adherence rate >= 75% (>= 18 hours/day) over a 4-week cycle (28 days) will be strongly encouraged.

SUMMARY:
This is a Phase 2 study in subjects with WHO Grade III Anaplastic Astrocytoma (G3 astrocytoma) who had progressive disease during first or second line treatment and who have not previously received any BEV or any experimental agents.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective will be to determine the efficacy of NOVOTTF-200A in recurrent anaplastic astrocytoma patients (6-month progression-free survival)

Secondary Objectives:

* To evaluate the safety of NOVOTTF-200A in the subject population.
* To evaluate efficacy of NOVOTTF-200A in the subject population.
* To see if the presence of ATRX, TERT promoter, IDH1 mutations and/or MGMT promoter methylation, confers a better response to NOVOTTF-200A.
* To determine if the treatment significantly modifies the patient's quality of life. Sponsor will use the Functional Assessment of Cancer Therapy (FACT) questionnaires:

  * FACT-Brain (FACT-Br)
  * FACT-Cognitive Function (FACT-Cog)

Exploratory Objectives:

* To determine if the presence of proneural or mesenchymal phenotype (Cytoscan analysis) confers a better response to NovoTTF.
* To determine if the in vitro sensitivity of the glioma cells derived from patient specimens before and after the NOVOTTF-200A treatment correlates with the patient's response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign and date an informed consent document before any study related assessments/procedures are conducted.
2. Males and females of age ≥18 years at the time of the signing of the informed consent document.
3. All subjects must have histologic evidence of G3 MG and radiographic evidence of recurrence or disease progression (defined as either a greater than 25% increase in the largest bi-dimensional product of enhancement, a new enhancing lesion or a significant increase in T2 FLAIR).
4. Subjects with archival tumor tissue suitable for genetic testing must give permission to access and test the tissue; subjects without archival tumor tissue are eligible.
5. No prior treatment with BEV or any anti-angiogenesis agents.
6. At least 4 weeks from surgical resection and 12 weeks from end of radiotherapy prior to enrollment in this study, unless relapse is confirmed by tumor biopsy or new lesion outside of radiation field, or if there are two MRIs confirming progressive disease that are 8 weeks apart.
7. All AEs resulting from prior chemotherapy, surgery or radiotherapy must have resolved to NCI-CTCAE (v. 4.03) Grade ≤1 (except for laboratory parameters outlined below).
8. Laboratory results within 7 days prior to NOVOTTF-200A administration (transfusions and/or growth factor support may be used at the discretion of the Investigator during Screening):

   * Hemoglobin ≥9 g/dL.
   * Absolute neutrophil count (ANC) ≥1.5 × 109/L.
   * Platelet count ≥100 × 109/L.
   * Serum bilirubin ≤1.5 × upper limit of normal (ULN) or ≤3 × ULN if Gilbert's disease is documented.
   * Aspartate transaminase (AST) ≤ 2.5 ULN.
   * Serum creatinine ≤1.5 × ULN.
9. Karnofsky Performance Status (KPS) score ≥70%.
10. Willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. The presence of 1p19q LOH which is diagnostic for anaplastic oligodendroglioma (AO).
2. Co-medication that may interfere with study results, e.g., immunosuppressive agents other than corticosteroids. (Steroid therapy for control of cerebral edema is allowed at the discretion of the investigator. Subjects should be on a stable dose of steroids for at least 1 week prior to study beginning.)
3. Chemotherapy administered within 4 weeks (6 weeks for an IV nitrosoureas and 12 weeks for an implanted nitrosoureas wafer) prior to Day 1 of study treatment.
4. Pregnancy or breastfeeding.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics & psychiatric illness/social situations that would limit adherence with study requirements, or disorders associated with significant immunocompromised state.
6. Known previous/current malignancy requiring treatment within ≤ 3 years except for cervical carcinoma in situ, squamous or basal cell skin carcinoma and superficial bladder carcinoma.
7. Any comorbid condition that confounds the ability to interpret data from the study as judged by the Investigator.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2025-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Bota, MD, Principal Investigator — UC Irvine Health
Locations (1):
- University of California, Irvine, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NOVOTTF-200A
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NOVOTTF-200A
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Showing no Evidence of Disease Progression Six Months After Initiating Treatment With the Device.
Description: The primary objective is to estimate the proportion of participants showing no evidence of disease progression six months after initiating treatment with the device. Assessment is per RANO (2010) criteria.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | NOVOTTF-200A
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Number of Participants Who Experience Any Adverse Events Who Received NOVOTTF-200A.
Description: All subjects will be evaluated for safety analysis if they receive NOVOTTF-200A. Safety and tolerability of NOVOTTF-200A treatment will be based on the incidence and severity of adverse events and toxicities. Toxicities will be assessed according to the "Common toxicity criteria (CTC), version 4.03". Refer to the Adverse Events (AEs) section for full list of reported AEs.
Time Frame: 1 year
Population: Refer to the Adverse Events (AEs) section for full list of reported AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | NOVOTTF-200A
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Does the Treatment Significantly Modify the Patient's Quality of Life?
Description: To determine if the treatment significantly modifies the patient's quality of life we will be using the Functional Assessment of Cancer Therapy (FACT) questionnaires that include the FACT-Brain (FACT-Br), and the FACT-Cognitive Function (FACT-Cog) questionnaires. These will be completed at baseline then every two cycles.
  Scores of FACT-COG and FACT-Br are combined below at baseline and last cycle of treatment. Scores of FACT-COG and FACT-Br are summed to obtain a total possible scale range of 0 to 272. FACT-Cog (using the Cognitive Impairments subscale) with a score range from 0-72 and FACT-Br with a score range from 0-200.
  A higher score, means a better quality of life.
Time Frame: Will be assessed at baseline and every two cycles (at the end of each even-numbered cycle of therapy) until treatment termination, an average of 24 months
Measure: Number; unit: score
Arm/Group | NOVOTTF-200A
Number analyzed (Participants) | 1
score
  Baseline | 239
  Last Cycle | 198

4. Secondary Outcome: Correlations With Established Molecular Markers (ATRX, and/or Mutation and MGMT Promoter Methylation
Description: To see if the presence of ATRX, TERT promoter, IDH1 mutations and/or MGMT promoter methylation, confers a better response to NOVOTTF-200A.
Time Frame: Assessed at screening.
Measure: Count of Participants; unit: Participants
Arm/Group | NOVOTTF-200A
Number analyzed (Participants) | 1
Participants
  ATRX | 0
  TERT promoter | 0
  IDH1 | 1
  MGMT | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected following initiation of treatment until 2 months after treatment termination, an average of 24 months.
Arm/Group | NOVOTTF-200A
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOVOTTF-200A (N=1)
Scalp Irritation (Skin and subcutaneous tissue disorders) | 1 (2)
Hearing Difference (Ear and labyrinth disorders) | 1 (1)
Flu-like Symptoms (General disorders) | 1
Conjunctivitis (Eye disorders) | 1
COVID-19 (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT03450850/Prot_SAP_000.pdf